CLINICAL TRIAL: NCT01288430
Title: A Phase 1, Open-Label, Multiple-Ascending-Dose Study of DS-2248, an Orally Bioavailable Heat Shock Protein 90 Inhibitor, in Subjects With Advanced Solid Tumors
Brief Title: A Study of DS-2248 in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was terminated as per Sponsor decision.
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo UK Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS2248-A-U101; 2011-002666-21 (EudraCT Number)
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Results first posted 2020-07-10 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Solid Tumors; Non-small Cell Lung Carcinoma
Keywords: Heat shock protein 90; Advanced solid tumors; Non-small cell lung carcinoma; Epidermal growth factor receptor; Tyrosine kinase inhibitor acquired resistance; Non-small cell lung carcinoma with acquired resistance to erlotinib, gefitinib, afatinib or others.
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DS-2248 (Experimental): Study Part 1: DS-2248 oral capsule(s) of increasing strength in a dose escalation study in subjects with advanced solid tumors, administered once daily in 21-day cycles, with no interruption between cycles if no unacceptable treatment-related toxicity or tumor progression is observed.
  Study Part 2: DS-2248 oral capsule(s) dose of 4.5 mg/m^2, in subjects with non-small cell lung cancer who have developed acquired resistance to epidermal growth factor receptor-tyrosine kinase inhibitors or whose tumors carry an ALK translocation and are resistant to ALK inhibitor therapy, administered once daily in 21 day-cycles, with no interruption between cycles if no unacceptable treatment-related toxicity or tumor progression are observed.
  Interventions: Drug: DS-2248

INTERVENTIONS:
Drug: DS-2248 — Oral capsules, of various strengths (1, 5 , 20 ,or 50 milligrams), once daily during 21-day cycles, until unacceptable treatment-related toxicity or tumor progression are observed.

SUMMARY:
This phase 1 clinical trial is intended to understand the safety and tolerability of a new anticancer drug in subjects with advanced solid tumors. The patients who qualify for the study will receive a once daily dose of the drug taken by mouth and will undergo several tests to measure the drug in the blood and to understand the safety, tolerability and any effect of the drug on the tumor. The antitumor effect of the drug is not known in human.

DETAILED DESCRIPTION:
The study will be conducted in two parts. Part 1 is a dose escalation study in which subjects in each cohort will be given increasing doses of the study drug until a maximum tolerated dose (MTD) or maximum administered dose (MAD) is determined as the recommended phase 2 dose (RP2D). The drug will be administered as oral capsules once daily in 21 day cycles, with no interruption between cycles if no unacceptable treatment-related toxicity or tumor progression are observed.

After determining the RP2D, Part 2 of the study, which is a dose expansion study will begin in which subjects with advanced non-small cell lung cancer who developed acquired resistance to epidermal growth factor receptor (EGFR)-tyrosine kinase inhibitors (TKI), erlotinib, gefitinib, afatinib (and others) or whose tumors carry an ALK translocation and are resistant to ALK inhibitor therapy, will be treated with DS-2248 at RP2D. The drug will be administered as oral capsules once daily in 21 day cycles, with no interruption between cycles if no unacceptable treatment-related toxicity or tumor progression are observed.

ELIGIBILITY:
Inclusion Criteria:

1. A pathologically documented advanced solid malignant tumor refractory to standard treatment or for which no standard treatment is available.
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
3. Have adequate bone marrow function, defined as:

   * Platelet count ≥100x10^9/L or more.
   * Hemoglobin (Hb) level ≥9.0 g/dL.
   * Absolute neutrophil count ≥1.5 x 10^9/L.
4. Have adequate renal function, defined as:

   - Creatinine clearance ≥60 mL/min, as calculated using the modified Cockcroft-Gault equation AND creatinine ≤1.5 times upper limit of normal(ULN).
5. Have adequate hepatic function, defined as:

   * Aspartate aminotransferase (AST) levels ≤3 times ULN (if liver metastases are present, ≤5x ULN)
   * Alanine aminotransferase (ALT) levels ≤3x ULN (if liver metastases are present, ≤5x ULN
   * Bilirubin ≤1.5x ULN
6. Have adequate blood clotting function, defined as:

   - Prothrombin time and activated partial thromboplastin time ≤1.5x ULN
7. Participants should be able to provide written informed consent, comply with protocol visits and procedures, be able to take oral medication, and not have any active infection or chronic co-morbidity that would interfere with therapy.
8. Participants (male and female) of childbearing/reproductive potential must agree to use double-barrier contraceptive measures or avoid intercourse during the study and for 90 days after the last dose of study drug. If female and of childbearing potential, must have a negative result of a pregnancy test (serum or urine)within 72 hours prior to initiating study treatment. Surgically sterile individuals and postmenopausal females are considered not having child-bearing potential.
9. Participants must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an Institutional Review Board approved informed consent form (including Health Insurance Portability and Accountability Act authorization, if applicable) before performance of any study-specific procedures or tests.
10. Participants must be willing to provide pre-existing diagnostic or resected tumor samples, such as formalin-fixed paraffin-embedded sections, if available. Providing fresh pre-treatment tumor biopsy is optional for participants in dose escalation cohorts and in dose expansion Stage 1. Post-treatment biopsies are optional for all the participants in the study (dose escalation and dose expansion cohorts).

Additional Inclusion Criteria for Part 2 (Dose Expansion)

1. Pathologically documented stage IIIB/IV non-small cell lung cancer.
2. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) criteria, Version 1.1.
3. Participants must meet 1 of the following 3 criteria in order to be included in Part 2:

   1. Acquired resistance to reversible Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitor (EGFR-TKI), which should meet the following criteria:

      * Previous treatment with single-agent therapy (erlotinib, gefitinib, afatinib or others).
      * Either of the following: A tumor that harbors an EGFR mutation known to be associated with drug sensitivity (i.e., G719X, exon 19 deletion, L858R, L861Q) -OR- Prior objective clinical benefit from EGFR-TKI, as evidenced by complete response (CR), partial response (PR), or stable disease (SD) ≥6 months as defined by RECIST or World Health Organization criteria.
      * Systemic progression of disease as defined by RECIST or World Health Organization criteria while treatment with gefitinib, erlotinib, afatinib or others.
      * No intervening therapy other than EGFR-TKIs (erlotinib, gefitinib, afatinib or others) after progression on an EGFR-TKI.
      * Pre-treatment biopsy (performed via bronchoscopy or imaging guidance) for molecular testing of the tumor is desired but not mandatory for enrollment in Stage 1. However, pre-treatment biopsy within 21 days prior to the first day of treatment is required for enrollment in Stage 2.
   2. Presence of ALK fusion gene in the tumor demonstrated by fluorescence in situ hybridization (FISH) and the participant has acquired resistance to ALK inhibitor therapy.

Exclusion Criteria:

1. History of second malignancies or primary central nervous system malignancies, except adequately treated non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated, with no evidence of disease for ≥3 years.
2. Gastrointestinal diseases that could affect the absorption of DS-2248.
3. Subjects with peptic ulcer disease requiring on-going treatment with pH-modifiers
4. Subjects with history of inflammatory bowel disease.
5. Subjects with retinal or uveal diseases including macular degeneration with central vision loss, retinal detachment, diabetic retinopathy, and uveitis.
6. Recipient of a stem cell or bone marrow transplant.
7. Has a concomitant medical condition that would increase the risk of toxicity, in the opinion of the Investigator or Sponsor.
8. Clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with steroids may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 4 weeks must have elapsed between the end of whole brain radiotherapy and study enrollment (2 weeks for stereotactic radiotherapy).
9. Has unresolved toxicities from previous anti-cancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0, Grade ≤1 or baseline. Subjects with chronic Grade 2 toxicities may be eligible per the discretion of the Investigator or Sponsor (e.g., Grade 2 chemotherapy-induced neuropathy).
10. Systemic treatment with anticancer therapy, antibody-based therapy, retinoid therapy, or hormonal therapy (except megestrol acetate as supportive care) within 3 weeks before study drug treatment; or treatment with nitrosoureas or mitomycin C within 6 weeks before study drug treatment; or treatment with small-molecule Tyrosine Kinase Inhibitors within 7 days for erlotinib and afatinib and 10 days for gefitinib before study drug treatment. Previous and concurrent use of hormone replacement therapy, the use of gonadotropin-releasing hormone modulators for prostate cancer, and the use of somatostatin analogs for neuroendocrine tumors are permitted.
11. Therapeutic radiation therapy or major surgery within 4 weeks before study drug treatment or palliative radiation therapy within 2 weeks before study drug treatment.
12. Participation in a clinical drug study within 3 weeks for small-molecule TKIs before study drug treatment, or current participation in other investigational procedures.
13. Concomitant treatment with potent inducers or potent inhibitors of cytochrome P450 3A4 (CYP3A4).
14. Concomitant treatment with a medication known to cause renal tubular damage or reduce renal perfusion at the dose administered, including aminoglycosides, amphotericin B, pentamidine, nonsteroidal anti-inflammatory drugs, and zoledronate.
15. Corrected QT interval (QTc by Bazett's formula) prolongation at rest, where the mean QTc interval is >450 msec based on triplicate ECG.
16. Pregnant or breastfeeding.
17. Substance abuse or medical, psychological, or social conditions that may, in the opinion of the Investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
18. Less than 1 week since using systemically acting drugs that increase gastric pH, such as H2-blockers and proton pump inhibitors. Antacids should be avoided within 48 hours of the first dose of DS-2248.
19. Use of St. John's Wort (hypericin) is not permitted for 30 days before and during the study. Foods or beverages containing grapefruit should be avoided within 48 hours before and during the study.

Additional Exclusion Criteria for Part 2 (Dose Expansion)

1. Prior treatment with Hsp90 inhibitors
2. Intervening therapy after progression on an EGFR-TKI (erlotinib, gefitinib, afatinib or others), unless re-treated with EGFR-TKI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03-29 (Actual); Primary Completion 2014-02-13 (Actual); Study Completion 2014-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (9):
- United States (9):
  - Duarte, California
  - Loma Linda, California
  - Orange, California
  - Orlando, Florida
  - Indianapolis, Indiana
  - Detroit, Michigan
  - Portland, Oregon
  - San Antonio, Texas
  - Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 participants who met all inclusion and no exclusion criteria were enrolled in the study.
Pre-assignment Details: Part 1: Dose escalation began with an accelerated titration design, with a starting dose of DS-2248 0.6 mg/m^2 once daily. Part 2: Dose expansion was assessed in participants with Stage IIIB/IV non-small cell lung cancer with resistance to epidermal growth factor receptor tyrosine kinase inhibitor or ALK inhibitor therapy.
Groups:
- Part 1, Cohort 1: DS-2248 0.6 mg/m^2: Participants who received oral DS-2248 0.6 mg/m^2 once daily.
- Part 1, Cohort 2: DS-2248 1.2 mg/m^2: Participants who received oral DS-2248 1.2 mg/m^2 once daily.
- Part 1, Cohort 3: DS-2248 1.8 mg/m^2: Participants who received oral DS-2248 1.8 mg/m^2 once daily.
- Part 1, Cohort 4: DS-2248 2.7 mg/m^2: Participants who received oral DS-2248 2.7 mg/m^2 once daily.
- Part 1, Cohort 5: DS-2248 3.5 mg/m^2: Participants who received oral DS-2248 3.5 mg/m^2 once daily.
- Part 1, Cohort 6: DS-2248 4.5 mg/m^2: Participants who received oral DS-2248 4.5 mg/m^2 once daily.
- Part 1, Cohort 7: DS-2248 5.85 mg/m^2: Participants who received oral DS-2248 5.85 mg/m^2 once daily.
- Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2: Participants who were epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI)-resistant and received oral 4.5 mg/m^2 once daily.
- Part 2, ALK-resistant: DS-2248 4.5 mg/m^2: Participants who were ALK-inhibitor resistant and received oral 4.5 mg/m^2 once daily.
- Part 2, ALK-naive: DS-2248 4.5 mg/m^2: Participants who were ALK treatment naive and received oral 4.5 mg/m^2 once daily.
Period: Part 1
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2
Started (Only participants enrolled in Pt 1 are reported in this section.) | 2 | 3 | 5 | 7 | 3 | 6 | 7 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 3 | 5 | 7 | 3 | 6 | 7 | 0 | 0 | 0
Not completed — Progressive disease | 2 | 1 | 1 | 6 | 2 | 4 | 2 | 0 | 0 | 0
Not completed — Clinical disease progression | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Not completed — Death due to disease progression | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Other | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2
Started (Only participants enrolled in Pt 2 are reported in this section.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 3
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 7 | 2
Not completed — Clinical disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographics and baseline characteristics were assessed in the Enrolled Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2 | Total
Number analyzed (Participants) | 2 | 3 | 5 | 7 | 3 | 6 | 7 | 12 | 12 | 3 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 3 | 5 | 2 | 6 | 4 | 7 | 8 | 3 | 40
  >=65 years | 2 | 1 | 2 | 2 | 1 | 0 | 3 | 5 | 4 | 0 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.0 (0.0) | 58.7 (16.6) | 61.0 (10.8) | 60.1 (11.9) | 53.0 (17.4) | 49.8 (11.6) | 61.4 (12.9) | 58.8 (11.2) | 59.8 (11.8) | 51.7 (2.5) | 58.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 4 | 1 | 2 | 2 | 6 | 5 | 2 | 29
  Male | 1 | 1 | 1 | 3 | 2 | 4 | 5 | 6 | 7 | 1 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
  White | 2 | 2 | 5 | 7 | 3 | 5 | 6 | 9 | 8 | 3 | 50
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5 | 7 | 3 | 6 | 7 | 12 | 12 | 3 | 60

OUTCOME MEASURES:

1. Primary Outcome: Summary of Objective Response Rate Following Oral Administration of DS-2248 in Participants With Advanced Solid Tumors
Description: Objective response rate was defined as the sum of complete response (CR) and partial response (PR) rates. CR was defined as a disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline up to disease progression, discontinuation of study, or death, up to 2 years 11 months
Population: Objective response rate was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2
Number analyzed (Participants) | 2 | 3 | 3 | 5 | 2 | 6 | 4 | 10 | 9 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Summary of Best Overall Response Rate Following Oral Administration of DS-2248 in Participants With Advanced Solid Tumors
Description: Complete response (CR) was defined as a disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to <10 mm. Partial response (PR) was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease (PD) was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. Stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Objective response rate (ORR) was defined as the sum of CR and PR rates.
Time Frame: Baseline up to disease progression, discontinuation of study, or death, up to 2 years 11 months
Population: Best overall response was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2
Number analyzed (Participants) | 2 | 3 | 3 | 5 | 2 | 6 | 4 | 10 | 9 | 2
Participants
  Confirmed CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Confirmed PR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable disease | 1 | 1 | 3 | 0 | 0 | 2 | 2 | 4 | 2 | 1
  Progressive disease | 1 | 1 | 0 | 5 | 2 | 3 | 2 | 6 | 7 | 1
  Non-evaluable | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

3. Secondary Outcome: Summary of Disease Control Rate Following Oral Administration of DS-2248 in Participants With Advanced Solid Tumors
Description: Disease control rate (DCR) was defined as the sum of complete response (CR) and partial response (PR) rates, and stable disease (SD) rate for a minimum of 12 weeks. Complete response (CR) was defined as a disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to <10 mm. Partial response (PR) was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (at least a 20% increase in the sum of diameters of target lesions), taking as reference the smallest sum diameters while on study.
Time Frame: Baseline up to disease progression, discontinuation of study, or death, up to 2 years 11 months
Population: Disease control rate was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2
Number analyzed (Participants) | 2 | 3 | 3 | 5 | 2 | 6 | 4 | 10 | 9 | 2
Participants | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 1

4. Secondary Outcome: Duration of Stable Disease Following Oral Administration of DS-2248 in Participants With Advanced Solid Tumors
Description: Duration of response measured from the time at which criteria were first met for complete (CR) or partial response (PR) until the first date that progressive disease (PD) was objectively documented. Participants who had not progressed at the data cut-off date were censored at their last evaluable tumor assessment date. Duration of stable disease (SD) measured from the date of enrollment until the first date that criteria for disease progression were met. The minimum time interval for the duration of SD was 6 weeks. Participants who had not progressed at the data cut-off date were censored at their last evaluable tumor assessment date.
Time Frame: Baseline up to disease progression, discontinuation of study, or death, up to 2 years 11 months
Population: Duration of stable disease was assessed in participants in which data were available in the Full Analysis Set.
Measure: Median (Full Range); unit: weeks
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2
Number analyzed (Participants) | 1 | 1 | 3 | 0 | 0 | 2 | 2 | 4 | 2 | 1
weeks | 15.00 [15.0 to 15.0] | 7.9 [7.9 to 7.9] | 13.29 [7.4 to 32.7] |  |  | 9.50 [6.4 to 12.6] | 6.64 [6.6 to 6.7] | 12.86 [7.0 to 14.3] | 10.57 [7.1 to 14.0] | 13.1 [13.1 to 13.1]

5. Secondary Outcome: Summary of Progression-free Survival Following Oral Administration of DS-2248 in Participants With Advanced Solid Tumors
Description: Progression-free survival (PFS) defined as the time from the date of enrollment to the earlier of the dates of the first objective documentation of radiographic disease progression (as per RECIST V1.1) or death due to any cause. Participants who were alive with no objective documentation of (radiographic) disease progression by the data cut-off date were censored at the date of their last evaluable tumor assessment. Participants who were lost to follow-up or withdrew early from the study with no documented disease progression were censored at the last evaluable tumor assessment.
Time Frame: Baseline up to disease progression, discontinuation of study, or death, up to 2 years 11 months
Population: Progression-free survival was assessed in the Full Analysis Set.
Measure: Median (Full Range); unit: weeks
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2
Number analyzed (Participants) | 2 | 3 | 3 | 5 | 2 | 6 | 4 | 10 | 9 | 2
weeks | 10.93 [6.9 to 15.0] | 5.71 [5.1 to 7.9] | 13.29 [7.4 to 32.7] | 7.00 [5.6 to 8.1] | 5.64 [4.0 to 7.3] | 6.00 [5.0 to 12.6] | 6.57 [6.4 to 6.7] | 7.21 [7.0 to 14.3] | 7.14 [5.6 to 14.0] | 10.00 [6.9 to 13.1]

6. Secondary Outcome: Summary of Pharmacokinetic Parameter Area Under the Concentration Versus Time Curve From Zero to Infinity Following Oral Administration of DS-2248 in Participants With Advanced Solid Tumors
Time Frame: Cycle 1, Day 1 predose, 0.5, 1, 2, 3, 4, 6, and 8 h postdose; Cycle 1, Day 2 and Day 15; Cycle 1, Day 8 predose, 1 and 6 h postdose; Cycle 2 and 3, Day 1, 8, and 15
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set for which data were available.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2
Number analyzed (Participants) | 1 | 3 | 3 | 1 | 1 | 5 | 3 | 9 | 5 | 1
ng*h/mL | 76.47 | 122.56 (60.78) | 186.16 (102.20) | 362.31 | 356.01 | 675.57 (478.25) | 837.50 (606.70) | 501.21 (161.80) | 645.62 (257.30) | 459.96

7. Secondary Outcome: Summary of Pharmacokinetic Parameter Maximum Concentration Following Oral Administration of DS-2248 in Participants With Advanced Solid Tumors
Time Frame: as for outcome 6
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set for which data were available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2
Number analyzed (Participants) | 2 | 3 | 5 | 7 | 3 | 6 | 7 | 12 | 12 | 3
ng/mL | 6.46 (1.54) | 14.69 (7.37) | 25.60 (9.62) | 63.27 (31.02) | 71.30 (37.99) | 77.15 (32.17) | 126.61 (67.60) | 82.56 (34.22) | 81.45 (53.71) | 84.97 (34.16)

8. Secondary Outcome: Summary of Pharmacokinetic Parameter Time at Maximum Concentration Following Oral Administration of DS-2248 in Participants With Advanced Solid Tumors
Time Frame: as for outcome 6
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set for which data were available.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2
Number analyzed (Participants) | 2 | 3 | 5 | 7 | 3 | 6 | 7 | 12 | 12 | 3
hours | 2.0 (1.4) | 1.7 (0.6) | 1.1 (0.6) | 1.5 (0.9) | 1.2 (0.8) | 2.3 (1.0) | 2.1 (0.7) | 1.8 (0.9) | 1.6 (0.9) | 2.0 (1.1)

9. Secondary Outcome: Summary of Pharmacokinetic Parameter Terminal Half-life Following Oral Administration of DS-2248 in Participants With Advanced Solid Tumors
Time Frame: as for outcome 6
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set for which data were available.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2
Number analyzed (Participants) | 1 | 3 | 3 | 1 | 1 | 5 | 3 | 9 | 5 | 1
hours | 9.58 | 7.81 (1.75) | 8.11 (1.79) | 10.78 | 8.57 | 8.62 (1.21) | 10.05 (0.73) | 9.94 (0.93) | 9.23 (0.55) | 6.76

10. Secondary Outcome: Summary of Pharmacokinetic Parameter Total Body Clearance Following Oral Administration of DS-2248 in Participants With Advanced Solid Tumors
Time Frame: as for outcome 6
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set for which data were available.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2
Number analyzed (Participants) | 1 | 3 | 3 | 1 | 1 | 5 | 3 | 9 | 5 | 1
L/h | 0.01 | 0.02 (0.01) | 0.01 (0.00) | 0.01 | 0.01 | 0.02 (0.01) | 0.02 (0.01) | 0.02 (0.00) | 0.01 (0.00) | 0.02

11. Secondary Outcome: Summary of Drug Related Treatment Emergent Adverse Events Following Oral Administration of DS-2248 in Participants With Advanced Solid Tumors
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event that emerges during treatment, having been absent at pre-treatment; or reemerges during treatment, having been present at baseline but stopped prior to treatment; or worsens in severity after starting treatment relative to the pre-treatment state, when the AE is continuous. A DS-2248-related TEAE is an TEAE that is related to DS-2248 in the relationship.
Time Frame: Baseline up to 30 days post last dose, up to 2 years 11 months
Population: Treatment-emergent adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Total - Part 1: All participants who received oral DS-2248 in Part 1.
- Total - Part 2: All participants who received oral DS-2248 in Part 2.
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Total - Part 1 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2 | Total - Part 2
Number analyzed (Participants) | 2 | 3 | 5 | 7 | 3 | 6 | 7 | 33 | 12 | 12 | 3 | 27
Participants
  Drug-related TEAEs | 1 | 0 | 4 | 5 | 1 | 4 | 6 | 21 | 7 | 9 | 2 | 18
  Blood and Lymphatic Disorders | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 4
  Anaemia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 4
  Thrombocytopenia | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Lymphopenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Cardiac Disorders | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Tachycardia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Eye Disorders | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 5
  Retinal haemorrhage | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Dry eye | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Photopsia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Vision blurred | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Vitreous floaters | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Gastrointestinal Disorders | 0 | 0 | 1 | 3 | 1 | 1 | 3 | 9 | 3 | 4 | 2 | 9
  Abdominal distension | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  Anorectal discomfort | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Constipation | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 1
  Diarrhoea | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 4
  Dyspepsia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Flatulence | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Nausea | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 4
  Vomiting | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 2
  Abdominal pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Gastrooesophageal reflux disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Paraesthesia oral | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  General Disorders & Administration Site Conditions | 0 | 0 | 3 | 1 | 0 | 2 | 2 | 8 | 3 | 3 | 1 | 7
  Fatigue | 0 | 0 | 3 | 1 | 0 | 2 | 2 | 8 | 3 | 2 | 1 | 6
  Oedema peripheral | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Irritability | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Immune System Disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Hypersensitivity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Investigations | 0 | 0 | 1 | 1 | 1 | 2 | 4 | 9 | 3 | 3 | 1 | 7
  Alanine aminotransferase increase | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1
  Aspartate aminotransferase increased | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0
  Blood alkaline phosphatase increased | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1
  Blood creatinine increased | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 5 | 1 | 0 | 0 | 1
  Blood urea increased | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Blood uric acid increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Blood phosphorus increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Weight decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Weight increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Metabolism and Nutrition Disorders | 1 | 0 | 1 | 2 | 0 | 2 | 2 | 8 | 3 | 1 | 2 | 6
  Decreased appetite | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 4 | 1 | 0 | 2 | 3
  Dehydration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Hyperglycaemia | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hyperphosphataemia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Hyperuricaemia | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Hypoalbuminaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Hypokalaemia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
  Musculoskeletal and Connective Tissue Disorders | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 3
  Arthralgia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Muscular weakness | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
  Musculoskeletal pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Myalgia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Nervous System Disorders | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 6 | 1 | 9
  Dizziness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
  Dysgeusia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 5 | 0 | 5
  Headache | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Nystagmus | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Restless legs syndrome | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Renal and Urinary Disorders | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Proteinuria | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Renal failure acute | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Respiratory, Thoracic, and Mediastinal Disorders | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Dyspnoea | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Reproductive System and Breast Disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Breast tenderness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Skin and Subcutaneous Tissue Disorders | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 4
  Dry skin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Hyperhidrosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Onychoclasis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Pruritus | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from baseline up to 30 days post last dose, up to 2 years 11 months.
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event (AE) that emerges during treatment, having been absent at pre-treatment; or reemerges during treatment, having been present at baseline but stopped prior to treatment; or worsens in severity after starting treatment relative to the pre-treatment state, when the AE is continuous.
Arm/Group | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 | Part 2, ALK-naive: DS-2248 4.5 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/5 | 0/7 | 1/3 | 0/6 | 0/7 | 0/12 | 0/12 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/3 | 2/5 | 3/7 | 1/3 | 1/6 | 1/7 | 1/12 | 0/12 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 5/5 | 7/7 | 3/3 | 6/6 | 7/7 | 12/12 | 10/12 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 (N=2) | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 (N=3) | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 (N=5) | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 (N=7) | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 (N=3) | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 (N=6) | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 (N=7) | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 (N=12) | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 (N=12) | Part 2, ALK-naive: DS-2248 4.5 mg/m^2 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device occlusion (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, Cohort 1: DS-2248 0.6 mg/m^2 (N=2) | Part 1, Cohort 2: DS-2248 1.2 mg/m^2 (N=3) | Part 1, Cohort 3: DS-2248 1.8 mg/m^2 (N=5) | Part 1, Cohort 4: DS-2248 2.7 mg/m^2 (N=7) | Part 1, Cohort 5: DS-2248 3.5 mg/m^2 (N=3) | Part 1, Cohort 6: DS-2248 4.5 mg/m^2 (N=6) | Part 1, Cohort 7: DS-2248 5.85 mg/m^2 (N=7) | Part 2, EGFR TKI-resistant: DS-2248 4.5 mg/m^2 (N=12) | Part 2, ALK-resistant: DS-2248 4.5 mg/m^2 (N=12) | Part 2, ALK-naive: DS-2248 4.5 mg/m^2 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 1 | 2 | 1 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 2 | 1
Fatigue (General disorders) | 1 | 1 | 3 | 4 | 2 | 4 | 4 | 5 | 3 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 2 | 1 | 3 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 4 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 2 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 4 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 2 | 1 | 1 | 4 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No